CLINICAL TRIAL: NCT01261078
Title: The Bupivacaine Dose Sparing Effect of Intrathecal Epinephrine for Spinal Anesthesia in Total Knee Replacement Arthroplasty
Brief Title: The Bupivacaine Dose Sparing Effect of Intrathecal Epinephrine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul Medical Center (Other)
Responsible Party: Won Ho Kim M.D. Faculty anesthesiologist, Seoul Meducal Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SMC-2010-12-05
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2010-12

CONDITIONS: Spinal Anesthesia
Keywords: intrathecal epinephrine; duration of anesthesia; quality of anesthesia; intrathecal fentanyl
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): 8 mg bupivacaine only
  Interventions: Drug: Placebo
- Epi 25 (Active Comparator): 8 mg of bupivacaine mixed with 25 mcg of epinephrine
  Interventions: Drug: epinephrine 25
- Epi 50 (Active Comparator): 8 mg of bupivacaine mixed with 50 mcg of epinephrine
  Interventions: Drug: Epinephrine 50
- Epi 100 (Active Comparator): 8 mg of bupivacaine mixed with 0.1 mg of epinephrine
  Interventions: Drug: epinephrine 100
- Epi 200 (Active Comparator): intrathecal bupivacaine 8 mg with 200 mcg of epinephrine
  Interventions: Drug: Epi 200

INTERVENTIONS:
Drug: Placebo — intrathecal 8 mg of bupivacaine only
  Other Names: Epinephrine
  Arms: Placebo
Drug: epinephrine 25 — intrathecal 8 mg of bupivacaine mixed with 25 mcg of epinephrine
  Other Names: Epinephrine
  Arms: Epi 25
Drug: Epinephrine 50 — intrathecal 8 mg of bupivacaine mixed with 50 mcg of epinephrine
  Other Names: Epinephrine
  Arms: Epi 50
Drug: epinephrine 100 — intrathecal 8 mg of bupivacaine mixed with 0.1 mg of epinephrine
  Other Names: Epinephrine
  Arms: Epi 100
Drug: Epi 200 — intrathecal bupivacaine 8 mg with 200 mcg of epinephrine
  Other Names: epinephrine
  Arms: Epi 200

SUMMARY:
Intrathecal epinephrine has been known to increase the duration of spinal anesthesia, or increase the quality of anesthesia. However, there is still a controversy, and the mechanism of epinephrine is recently suggested as a modulator of pain information in the spinal cord. Therefore, the investigators try to investigate the dose sparing effect of intrathecal epinephrine for spinal anesthesia with bupivacaine.

DETAILED DESCRIPTION:
For patient undergoing total knee replacement arthroplasty, patients injected intrathecally with bupivacaine 8 mg were compared with those with bupivacaine 8 mg with 25 mcg of epinephrine, bupivacaine 8 mg with 50 mcg of epinephrine, and those with bupivacaine 8 mg with 100 mcg of epinephrine. The investigators compared the characteristics of spinal anesthesia including the quality and complication of spinal anesthesia. The researchers investigated whether intrathecal dose of epinephrine can reduce bupivacaine requirement and this effect is dependent on the dose of epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing total knee replacement arthroplasty

Exclusion Criteria:

* patient with cardiac or pulmonary disease (ASA class III or more)
* patient undergone previous spine surgery
* patient undergoing revised knee replacement

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
the sensory level of spinal anesthesia, the quality of intraoperative analgesia | every 15 minutes
  at 2, 5, 10, 20, and 30 min after the spinal injection and every 15 minutes thereafter until complete regression of spinal anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, M.D., Principal Investigator — Seoul Medical Center
Locations (1):
- Seoul Medical Center, Seoul, South Korea